CLINICAL TRIAL: NCT02956005
Title: Envarsus XR in African American Renal Transplant Recipients
Acronym: EXR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IIS - PI left the institution. Subjects just followed to study completion
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXR1
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2016-11

CONDITIONS: Renal Transplant Recipients
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Envarsus (Other): Open Label; Envarsus XR started at the time of transplant. Initial dosing of 0.17mg/kg. Target trough level of 8-10 ng/mL
  Interventions: Drug: ENVARSUS®

INTERVENTIONS:
Drug: ENVARSUS® — ENVARSUS XR is a form of the anti-rejection drug, tacrolimus, for people who have had a kidney transplant
  Other Names: Extended Release Tacrolimus

SUMMARY:
The purpose of this study is to collect data prospectively on African American patients who are taking the immunosuppressant Envarsus post kidney transplant. We are looking to see if African American renal transplant recipients that receive Envarsus will have less tubular injury and calcenurin inhibitor toxicity compared with patients that receive tacrolimus IR.

African americans have the higher rates of CYP3A5 which is associated with the need of higher tacrolimus dose to achieve an adequate level and this many times is associated with signs and symptoms of tacrolimus toxicity such as tremors, headaches and neuropathies.

The retrospective cohort will be African American patients that will be matched by age, gender, type of kidney transplant (living vs deceased) and level of sensitization

ELIGIBILITY:
Inclusion Criteria:

1. African American race
2. Adult renal transplant recipients (>18 y/o)
3. Previous adverse reaction or contraindication to the use of tacrolimus

Exclusion Criteria:

1. Non African American race
2. Less than 18 y/o (pediatric patients)
3. Recipients of liver and small bowel transplants
4. Adverse reaction to tacrolimus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Envarsus
Started | 18
Completed | 2
Not Completed | 16
Not completed — Not eligible | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 12

BASELINE CHARACTERISTICS:
Arm/Group | Envarsus
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint is to Determine the Rate of Calcineurin Inhibitor Toxicity as Measured by Surveillance Kidney Biopsies.
Description: Data not collected - study terminated prematurely when PI left institution.
Time Frame: 1 year
Population: Analysis not completed - PI left institution
Arm/Group | Envarsus
Number analyzed (Participants) | 0

2. Secondary Outcome: Renal Function After Transplantation
Description: Data not collected - study terminated prematurely when PI left institution.
Time Frame: 1 year
Population: PI left institution - Analysis not completed
Arm/Group | Envarsus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the patient received the first dose until study completion (12 months) or withdrawal, whichever occurred first
Description: No difference from clinicaltrials.gov definition
Arm/Group | Envarsus
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Envarsus (N=18)
Acute Kidney Injury (Injury, poisoning and procedural complications) | 4 (4)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension Urgency (Vascular disorders) | 1 (1)
Muscle Tremor (Musculoskeletal and connective tissue disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delayed Graft Function (Renal and urinary disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liver Resection of HCC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute Kidney Failure (Renal and urinary disorders) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Flu (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Envarsus (N=18)
Hypertension (Vascular disorders) | 7 (7)
Worsening Hypertension (Vascular disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Worsening Anemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Delayed Graft Function (Renal and urinary disorders) | 1 (1)
Slow Graft Function (Renal and urinary disorders) | 6 (6)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 2 (2)
Coronary Artery Disease (Vascular disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 (3)
Diabetes (Endocrine disorders) | 2 (2)
CMV (Infections and infestations) | 1 (1)
BK Viremia (Infections and infestations) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (2)
Incisional Pain (Injury, poisoning and procedural complications) | 4 (4)
Weakness/Fatiugue (General disorders) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Secondary Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2)
Nausea/Emesis (Gastrointestinal disorders) | 6 (6)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Genital Ulcer (Reproductive system and breast disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neurological Symptoms (Nervous system disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Hypercholesterolemia (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypovolemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 3 (3)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 5 (5)
Ileus (Gastrointestinal disorders) | 1 (1)
DSA (Immune system disorders) | 2 (2)
Elevated intra-operative blood pressure (Vascular disorders) | 1 (1)
Acute Kidney Injury (Injury, poisoning and procedural complications) | 1 (1)
Frequent Urination (Renal and urinary disorders) | 1 (1)
Burning after Urination (Renal and urinary disorders) | 1 (1)
Wound Tear (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Improper Wound Healing (Injury, poisoning and procedural complications) | 1 (1)
Elevated Creatinine (Investigations) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Transplant Adhesion (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
Hemolytic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Chronic Anticoagulation (Blood and lymphatic system disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (2)
HCV (Infections and infestations) | 1 (1)
Lack of appetite (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The PI of this study left the institution before the study was completed. Patients were followed until the completion of the study if applicable, but no study data analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT02956005/Prot_SAP_000.pdf